CLINICAL TRIAL: NCT01849302
Title: The Acute Effect of Beverages Varying in Macro-nutrient Content on Subjective Appetite Ratings and ad Libitum Energy Intake in Healthy Subjects
Brief Title: The Effect of Beverages Varying in Protein Quantity on Appetite and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anestis Dougkas, Postdoctoral Research Fellow, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/6
Record Dates: First submitted 2013-04-30; First posted 2013-05-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Appetite; Satiety hormones; Dietary Protein
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- High protein/ High fat beverage (Experimental): Beverage based on milk protein: 1.8 MJ, 40 E% Protein, 42 E% fat
  Acute effect of beverages varying in macronutrient content on appetite and energy intake
  Interventions: Dietary Supplement: Beverages varying in macronutrient content on appetite
- High protein/ Normal CHO beverage (Experimental): Beverage based on milk protein: 1.8 MJ, 40 E% Protein, 47 E% CHO
  Acute effect of beverages varying in macronutrient content on appetite and energy intake
  Interventions: Dietary Supplement: Beverages varying in macronutrient content on appetite
- Low protein/ High fat beverage (Experimental): Beverage based on milk protein: 1.8 MJ, 9 E% Protein, 63 E% fat
  Acute effect of beverages varying in macronutrient content on appetite and energy intake
  Interventions: Dietary Supplement: Beverages varying in macronutrient content on appetite
- Low protein/ High CHO beverage (Experimental): Beverage based on milk protein: 1.8 MJ, 9 E% Protein, 71 E% CHO
  Acute effect of beverages varying in macronutrient content on appetite and energy intake
  Interventions: Dietary Supplement: Beverages varying in macronutrient content on appetite
- Normal protein/ Normal CHO beverage 1 (Experimental): Beverage based on milk protein: 1.8 MJ, 24 E% Protein, 50 E% CHO
  Acute effect of beverages varying in macronutrient content on appetite and energy intake
  Interventions: Dietary Supplement: Beverages varying in macronutrient content on appetite
- Normal protein/Normal CHO beverage 2 (Experimental): Beverage based on milk protein: 1.8 MJ, 24 E% Protein, 50 E% CHO
  Acute effect of beverages varying in macronutrient content on appetite and energy intake
  Interventions: Dietary Supplement: Beverages varying in macronutrient content on appetite
- Normal protein/Normal CHO beverage 3 (Experimental): Beverage based on milk protein: 1.8 MJ, 24 E% Protein, 50 E% CHO
  Acute effect of beverages varying in macronutrient content on appetite and energy intake
  Interventions: Dietary Supplement: Beverages varying in macronutrient content on appetite

INTERVENTIONS:
Dietary Supplement: Beverages varying in macronutrient content on appetite — In this randomized, within-subject study, subjects are asked to consume 7 iso-energetic and iso-volumetric beverages as breakfast (20% of estimated energy requirements) with varying distribution of macronutrients. The objective is to identify the optimal protein quantity or macronutrient distribution on suppressing appetite.

SUMMARY:
Over the last decades, changes in the diet and lifestyle have led to overall energy imbalance becoming commonplace and the emergence of an obesity epidemic with more than 1.6 billion adults being overweight.

Consumption of foods that can affect appetite by increasing satiety could regulate the total energy intake and thus body weight. There is data suggesting that the macronutrient composition of the foods and especially protein content may have a potent role on satiety. However, it is difficult to pinpoint the optimum quantity needed to observe significant effects of protein on satiety.

The research project is dedicated to identify which food components [proteins, carbohydrates (CHO), fats] and the optimized protein quantity needed to accelerate satiation, suppress appetite and extend satiety until hunger appears again.

It is hypothesized that the consumption of protein-enriched meals will induce a reduction in hunger through the impact on gut hormones and peptides that are closely related to the short-term regulation of food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Age range 18-50 years
* Normal weight and overweight people as classified by BMI:22-27.9 kg/m2 (inclusive).
* Weight stable (within 3 kg) two months prior to study inclusion
* Understanding English well and feeling comfortable speaking it

Exclusion Criteria:

* Dietary protein consumption >25% energy from protein
* Had surgery in the previous 12 months
* Have suffered a myocardial infarction or stroke at any time
* Suffer from any blood-clotting disorder or prescription of any medication affecting blood clotting
* Suffer from any metabolic disorders (e.g. diabetes, metabolic syndrome or hypertension)
* Any requirement to take long-term medication, especially those active on the gastro-intestinal tract or for cardio-vascular disease
* Any dietary restrictions or recently/currently on a weight reducing diet
* Irregular eating patterns or not regularly consuming breakfast
* Food allergies (e.g. milk protein allergies) or intolerances (e.g. lactose)
* Use of medication which affects food intake or behaviour (e.g. anti-depressants)
* Use of medication likely to affect taste, smell or appetite
* Eating restraint based on the three Factor Eating Questionnaire
* Use of any protein supplements
* A history of alcohol or drug misuse (the average daily number of units of alcohol considered as acceptable is 2-3 units women; 3-4 units men
* Smoking
* Athletes in training (>10 h exercise/week)
* Female that is breast-feeding, pregnant, or if of child-bearing potential and are not using effective contraceptive precautions
* Involvement in a study involving an experimental drug/medication within 3 months prior to entry of this study
* Blood pressure > 160/90 mmHg
* Vegan or Vegetarian
* Glucose > 6 mmol/L
* Gamma glutamyl transferase > 1.9 μkat / L
* Alanine transaminase > 1.1 μkat / L
* Cholesterol > 6.5 mmol/L
* Triglycerides > 2.0 mmol/L

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in perceived appetite and satiety | Assessed every 30 min for 270 min after each of the seven beverages which are served at least one week apart (7 weeks)
  The appetite profile is assessed using validated Visual Analogue Scales (VAS) ratings (i.e hunger, fullness, desire to eat, prospective food consumption). The Questionnaires are performed electronically in personal laptops using the Adaptive Visual Analogue Scales (AVAS) software.

SECONDARY OUTCOMES:
Ad libitum energy intake | Energy intake is assessed 210 min after the 7 test beverages, which are served one week apart.
  Energy intake is assessed by ad libitum hot pasta meal provided 210 min after the test beverages, which are given as breakfast. Subjects are instructed to eat only until they feel comfortable satisfied and are given 25min to consume the meal. The total energy consumed is monitored
Changes from baseline in the postprandial concentration of satiety hormones | Assessed at 6 points in time over the morning of each of the 7 test days, which are separated by 1 week (7 weeks)
  Blood samples (2 ml) are collected at 0 min (fasted blood sample), 30, 60, 90, 150 and 205 min (i.e. total of 6 samples) over the morning on each test day (separated by 1 week) to quantify the plasma concentrations of circulating appetite regulating hormones. Protease inhibitors are added to the samples to reduce protein degradation. All samples are centrifuged at 4 C for 10 min at 2000 g after collection and are separated and stored in cryogenic vials at -80 C.
Hedonic ratings and palatability of the test beverages and meals | Assessed immediately after consumption of the 7 test beverages and pasta meal (7 weeks)
  The palatability and hedonic ratings are assessed using validated Visual Analogue Scales (VAS) ratings (i.e appearance, taste, overall palatability). The Questionnaires are performed electronically in personal laptops using the Adaptive Visual Analogue Scales (AVAS) software.
Changes from baseline in the postprandial concentration of glucose | Assessed at 7 points in time over the morning of each of the 7 test days, which are separated by 1 week (7 weeks)
  Capillary blood samples are collected by finger-prick at 0 min (fasted blood sample), 30, 45, 60, 90, 150 and 205 min (i.e. total of 7 samples) over the morning on each test day (separated by 1 week) to quantify the glucose concentration using HemoCue Glucose System.

CONTACTS AND LOCATIONS:
Overall Officials: Anestis Dougkas, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Applied Nutrition and Food Chemistry, Lund, Skåne County, Sweden

REFERENCES:
- [Derived] Dougkas A, Ostman E. Protein-Enriched Liquid Preloads Varying in Macronutrient Content Modulate Appetite and Appetite-Regulating Hormones in Healthy Adults. J Nutr. 2016 Mar;146(3):637-45. doi: 10.3945/jn.115.217224. Epub 2016 Jan 20. PMID 26791555